CLINICAL TRIAL: NCT04984876
Title: A 52 Week, Multi-center, Randomized, Double-blind Placebo-controlled Study to Assess the Clinical Efficacy and Safety of Ligelizumab (QGE031) in Decreasing the Sensitivity to Peanuts in Patients With Peanut Allergy
Brief Title: Efficacy and Safety of QGE031 (Ligelizumab) in Patients With Peanut Allergy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQGE031G12301; 2020-005339-56 (EudraCT Number); EMEA-001811-PIP03-20 (Other: EMA paediatric investigation plan number)
Record Dates: First submitted 2021-07-29; First posted 2021-08-02 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Allergy, Peanut
Keywords: Food allergy; Peanut allergy; Oral food challenge; IgE; ligelizumab
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity | interventions — ligelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ligelizumab 240 mg (Experimental): ligelizumab 240 mg subcutaneous injection for 52 weeks
  Interventions: Drug: ligelizumab
- ligelizumab 120 mg (Experimental): ligelizumab 120 mg subcutaneous injection for 52 weeks
  Interventions: Drug: ligelizumab
- Placebo 8 weeks and ligelizumab 120 mg (Experimental): Placebo subcutaneous injection for first 8 weeks and ligelizumab 120 mg subcutaneous injection for 44 weeks
  Interventions: Drug: ligelizumab; Drug: Placebo
- Placebo 16 weeks and ligelizumab 120 mg/240 mg (Experimental): Placebo subcutaneous injection for first 16 weeks and ligelizumab 120 mg OR 240 mg subcutaneous injection for 36 weeks
  Interventions: Drug: ligelizumab; Drug: Placebo
- Placebo 8 weeks and ligelizumab 240 mg (Experimental): Placebo subcutaneous injection for first 8 weeks and ligelizumab 240 mg subcutaneous injection for 44 weeks
  Interventions: Drug: ligelizumab; Drug: Placebo

INTERVENTIONS:
Drug: ligelizumab — Subcutaneous injection once every 4 weeks
Drug: Placebo — Subcutaneous injection once every 4 weeks
  Arms: Placebo 16 weeks and ligelizumab 120 mg/240 mg; Placebo 8 weeks and ligelizumab 120 mg; Placebo 8 weeks and ligelizumab 240 mg

SUMMARY:
This was a 52-week, Phase 3 multi-center, randomized, double-blind and placebo-controlled study to assess the safety and clinical efficacy of two dosing regimens of ligelizumab (240 mg and 120 mg) SC q4w (subcutaneous injection every 4 weeks) in participants with a medically confirmed diagnosis of Immunoglobulin E (IgE) mediated peanut allergy.

DETAILED DESCRIPTION:
Participants were randomized to ligelizumab 240 mg, ligelizumab 120 mg, or placebo (5 treatment arms, randomization ratio of 2:2:2:2:1) for the double-blind placebo-controlled treatment period (up to Week 12).

Participants initially assigned to the 8-week placebo arms received the first dose of blinded ligelizumab treatment at the Week 8 visit. Participants initially assigned to the 16-week placebo arm received the last dose of placebo before the Double Blind Placebo Controlled Food Challenge (DBPCFC) at Week 12 and the first dose of blinded ligelizumab treatment at the Week 16 visit.

At the start of the study, recruitment was restricted to 12-55-year-old participants. After approximately 60 adolescent participants (defined as 12-17 yrs of age) had completed all Week 12 assessments, an interim analysis (IA1) on Pharmacokinetics (PK) and selected Pharmacodynamics (PD) data (total IgE and basophil bound High affinity immunoglobulin E receptor 1 (FcƐRI)) was performed (safety was reviewed by a Data Monitoring Committee - DMC). Independent sponsor members who were responsible for PK/ PD data analysis and Modeling & Simulation were unblinded to the results of this interim analysis. The planned intent of this analysis was to confirm the dosing strategy for the youngest age group, 6-11 yrs and once the dose was to be confirmed, recruitment was supposed to be open for this age group. However, Novartis made a strategic decision to close recruitment in the study CQGE031G12301 and to terminate the study early, once all eligible participants in the study had completed week 12 assessments and the 16-week safety follow-up period. This decision was based on a blinded data review, which showed evidence of efficacy without the detection of any safety signal and that efficacy may be optimized with a different dosing regimen. Due to this decision, the final population size was 211, with only adolescent and adult participants (12 - 17yrs, and 18 - 55yrs) recruited.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent and/or assent (where applicable) was obtained prior to study participation. Participant (and parent/legal guardian) was able to understand and provide informed consent and assent, as applicable. If a minor participant providing assent reaches the age of legal majority (as defined by local law), he/she was re-consented (ICF) at the next study visit.
2. Male or female participants who were 6 to 55 yrs of age at the time of signing informed consent/assent.
3. Documented medical history of allergy to peanuts or peanut-containing foods.
4. Positive peanut-specific IgE (peanut sIgE), ≥ 0.35 kUA/L at Screening Visit 1.
5. Positive SPT for peanut allergen at Screening Visit 1. This is defined as the average diameter (longest diameter and mid-point orthogonal diameter) ≥ 4 mm wheal compared to the negative control.
6. A positive peanut DBPCFC at baseline (Screening Visit 2, Part 1 and Part 2 DBPCFC) defined as the occurrence of dose-limiting symptoms at a single dose ≤ 100 mg of peanut protein. Eligibility to proceed with the DBPCFC requires presence of all inclusion and absence of all exclusion criteria.
7. Participants must weigh ≥ 20 kg at Screening Visit 1.
8. Participants must be able to receive injections (study treatment), participate in the DBPCFC, and must be willing to continue avoiding exposure to peanuts and any other foods that they are allergic to throughout this study.

Key Exclusion Criteria:

1. History of hypersensitivity to ligelizumab or its excipients, or to other biologics (i.e., to murine, chimeric or human antibodies).
2. Hypersensitivity or intolerance to any of the matrix components used within the material for the oral food challenge.
3. History of severe or life-threatening hypersensitivity event needing an ICU (intensive care unit) admission or intubation within 60 days prior to baseline DBPCFC (Screening Visit 2).
4. Total IgE >2000 IU/mL at Screening Visit 1.
5. Participants with uncontrolled asthma (according to Global Initiative for Asthma (GINA) guidelines, GINA 2020) who meet any of the following criteria:

   * FEV1 <80% of participant's predicted normal value at Screening Visit 1
   * One hospitalization for asthma within 12 months prior to Screening Visit 1
6. Current or previous history of a mast cell disorder, including mastocytosis.
7. Platelets < 100'000/μL at Screening Visit 1.
8. Female participants not on oral contraception with a stable dose for a minimum of 3 months prior to taking study treatment.
9. Participants with evidence of helminthic parasitic infection as evidenced by stools being positive for a pathogenic organism according to local guidelines at Screening Visit 1 (before start of Screening Visit 2). If stool testing is positive for pathogenic organisms, the participant should not be randomized and should not be allowed to be rescreened.

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 211 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (29):
  - Allervie Clinical Research, Birmingham, Alabama
  - Allergy and Immunology Associates, Scottsdale, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Allergy and Asthma Associates of Santa Clara Vally Center, San Jose, California
  - Allergy and Asthma Clinical Research Inc, Walnut Creek, California
  - UCHealth Outpatient Pavilion, Aurora, Colorado
  - Asthma and Allergy Associates P C, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Ctr PC, Denver, Colorado
  - Univ of South Florida Asthma Allergy and Immunology CRU, Tampa, Florida
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Atlanta Allergy and Asthma Clinic, Marietta, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Family Allergy and Asthma, Louisville, Kentucky
  - Johns Hopkins Childrens Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Childrens Hospital, Boston, Massachusetts
  - University of Michigan Clinical Trials Office, Ann Arbor, Michigan
  - Respiratory Medicine Research Institute of Michigan, Ypsilanti, Michigan
  - UBMD Pediatrics, Buffalo, New York
  - Northwell Health, New York, New York
  - Mt Sinai Medical Center, New York, New York
  - University Of NC At Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Childrens Hospital MC, Cincinnati, Ohio
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Childrens Hospital, Houston, Texas
  - Seattle Allergy and Asthma Rsch, Seattle, Washington
- Australia (3):
  - Novartis Investigative Site, Brisbane, Queensland
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Canada (5):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Novartis Investigative Site, Odense, Denmark
- France (4):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
- Novartis Investigative Site, Padua, PD, Italy
- Japan (3):
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
- Novartis Investigative Site, Utrecht, Netherlands
- Spain (3):
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 56 centers in 10 countries worldwide
Groups:
- Placebo 16 Weeks and Ligelizumab 240 mg: Placebo subcutaneous injection for first 16 weeks and ligelizumab 240 mg subcutaneous injection for 36 weeks
- Placebo 16 Weeks and Ligelizumab 120 mg: Placebo subcutaneous injection for first 16 weeks and ligelizumab 120 mg subcutaneous injection for 36 weeks
Period: Overall Study
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo 16 Weeks and Ligelizumab 240 mg | Placebo 16 Weeks and Ligelizumab 120 mg
Started | 47 | 51 | 46 | 44 | 11 | 12
Randomized Analysis Set (RAS) (All randomized participants, regardless of whether or not they receive a dose of study drug) | 47 | 51 | 46 | 44 | 11 | 12
Full Analysis Set (FAS) (All participants who received at least one dose of study treatment. Mis-randomized patients (mis-randomized in IRT) will be excluded from FAS) | 47 | 51 | 46 | 44 | 11 | 12
Safety Set (SAF) (All participants who received at least one dose of study treatment whether or not being randomized) | 47 | 51 | 46 | 44 | 11 | 12
Completed | 44 | 40 | 41 | 37 | 8 | 11
Not Completed | 3 | 11 | 5 | 7 | 3 | 1
Not completed — Subject decision | 2 | 10 | 3 | 3 | 3 | 0
Not completed — Guardian decision | 0 | 1 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo 16 Weeks and Ligelizumab 240 mg | Placebo 16 Weeks and Ligelizumab 120 mg | Total
Number analyzed (Participants) | 47 | 51 | 46 | 44 | 11 | 12 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.5 (7.50) | 18.8 (6.27) | 18.7 (6.95) | 20.0 (7.75) | 17.4 (4.57) | 16.1 (3.58) | 18.9 (6.85)
Age, Customized [Count of Participants; unit: Participants]
  12 - 17 years | 27 | 29 | 25 | 24 | 6 | 8 | 119
  18 - 55 years | 20 | 22 | 21 | 20 | 5 | 4 | 92
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 19 | 20 | 3 | 6 | 98
  Male | 22 | 26 | 27 | 24 | 8 | 6 | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 10 | 2 | 1 | 2 | 2 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 1 | 2 | 0 | 0 | 12
  White | 31 | 36 | 42 | 39 | 7 | 10 | 165
  More than one race | 1 | 1 | 0 | 2 | 1 | 0 | 5
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 1 | 0 | 4
Time to diagnosis of peanut allergy [Mean (Standard Deviation); unit: Years] | 16.287 (7.9393) | 16.381 (6.9248) | 15.556 (7.5799) | 17.748 (7.8969) | 15.598 (5.3525) | 14.971 (3.5291) | 16.344 (7.2808)
Number of participants with at least one food allergy [Count of Participants; unit: Participants]
  1 food allergy | 12 | 15 | 13 | 11 | 5 | 3 | 59
  2 food allergies | 10 | 5 | 8 | 4 | 1 | 1 | 29
  3 food allergies | 5 | 5 | 2 | 5 | 3 | 1 | 21
  4 food allergies | 8 | 7 | 6 | 4 | 0 | 1 | 26
  5 food allergies | 0 | 4 | 4 | 3 | 1 | 2 | 14
  > 5 food allergies | 12 | 15 | 13 | 17 | 1 | 4 | 62
Peanut specific Immunoglobulin E (IgE) [Mean (Standard Deviation); unit: IU/mL] | 109.021 (147.9877) | 80.644 (117.6312) | 131.948 (189.7757) | 116.198 (128.9151) | 51.606 (48.6951) | 262.136 (543.7764) | 114.372 (191.3605)
Total Immunoglobulin E (IgE) [Mean (Standard Deviation); unit: IU/mL] | 524.35 (444.009) | 482.25 (478.047) | 455.38 (397.960) | 436.31 (335.113) | 325.15 (208.482) | 635.42 (535.099) | 476.81 (418.656)
MTD (maximum tolerated dose) of peanut protein (mg) - n (%) [Count of Participants; unit: Participants]
  < 1 mg | 2 | 5 | 2 | 2 | 1 | 0 | 12
  1 mg | 4 | 4 | 6 | 9 | 1 | 2 | 26
  3 mg | 14 | 14 | 11 | 11 | 1 | 1 | 52
  10 mg | 9 | 14 | 7 | 11 | 4 | 5 | 50
  30 mg | 18 | 14 | 20 | 11 | 4 | 4 | 71
Peanut Skin Prick Test (SPT) (undiluted): Size of mean wheal diameter [Mean (Standard Deviation); unit: mm] — Size of Mean wheal diameter (mm) = [(Mean of peanut wheal longest diameter + Mean of peanut wheal orthogonal diameter)/2]- average of the non-missing negative control diameters Population: Participants for which baseline data are not available are not counted.
  mm
    number analyzed (Participants) | 47 | 51 | 45 | 44 | 10 | 12 | 209
    (all) | 13.83 (5.720) | 14.61 (6.007) | 13.23 (6.414) | 16.82 (8.262) | 14.45 (4.845) | 12.17 (3.664) | 14.45 (6.508)
Peanut Skin Prick Test (SPT) (average across dilutions): Size of mean wheal diameter [Mean (Standard Deviation); unit: mm] — Size of Mean wheal diameter (mm) = [(Mean of peanut wheal longest diameter + Mean of peanut wheal orthogonal diameter)/2]- average of the non-missing negative control diameters. Range of dilutions (1:10 to 1:100,000). Population: Participants for which baseline data are not available are not counted.
  mm
    number analyzed (Participants) | 47 | 51 | 46 | 44 | 10 | 12 | 210
    (all) | 7.232 (2.8339) | 7.273 (2.7253) | 7.508 (2.7624) | 7.907 (2.8866) | 6.575 (2.3809) | 7.743 (2.3547) | 7.442 (2.7463)
Poly-sensitized to food [Count of Participants; unit: Participants] — Poly-sensitization is defined as specific Immunoglobulin E (sIgE) >=0.35kUA/L for a food allergen in the panel other than peanut.
  Participants
    Yes | 29 | 27 | 22 | 27 | 8 | 8 | 121
    No | 18 | 24 | 24 | 17 | 3 | 4 | 90
Poly-allergic to food [Count of Participants; unit: Participants] — Poly-allergic: Participants experiencing more than one food allergies in medical history.
  Participants
    Yes | 35 | 36 | 33 | 33 | 6 | 9 | 152
    No | 12 | 15 | 13 | 11 | 5 | 3 | 59
History of anaphylactic reaction to food [Count of Participants; unit: Participants]
  Yes | 32 | 36 | 29 | 32 | 9 | 8 | 146
  No | 14 | 15 | 16 | 12 | 2 | 4 | 63
  Unknown | 1 | 0 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Tolerated a Single Dose of >= 600 mg (1044 mg Cumulative Tolerated Dose) of Peanut Protein Without Dose-limiting Symptoms at Week 12
Description: Responder rate was defined as the percentage of participants tolerating a single dose of >= 600 mg (1044 mg cumulative tolerated dose) of peanut protein without dose-limiting symptoms during the double blind placebo controlled food challenge (DBPCFC) conducted at Week 12. The cumulative tolerated dose is the sum of the tolerated doses, not including the reactive dose. Dose-limiting symptoms indicate a true allergic reaction occurring during administration of a single dose of peanut protein at the DBPCFC that should preclude the administration of any further doses in the view of the investigator. Symptoms that require administration of any rescue medication were considered dose-limiting symptoms. Participants with treatment discontinuation or missing more than 1 doses of study drug prior to Week 12 due to reasons other than operational complications caused by public health emergency were considered non-responders.
Time Frame: Week 12
Population: Full Analysis Set (FAS). This outcome measure applies to ligelizumab 120 mg arm, ligelizumab 240 mg arm, and placebo 16-week to ligelizumab 120/240 mg arm (labelled as placebo for efficacy estimands).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo subcutaneous injection for first 16 weeks and ligelizumab 120 mg OR 240 mg subcutaneous injection for 36 weeks
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 47 | 51 | 23
Participants | 21 | 8 | 1
Statistical Analysis 1: Comparison: Ligelizumab 240 mg vs Placebo; Test type: Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 25.83, 95% CI 2-sided [4.34 to 506.78] — logistic regression model, including treatment, age subgroup (12 - 17 yrs, 18 - 55 yrs), region as fixed class effects, as well as and log-transformed baseline total IgE at screening and log-transformed MTD at screening DBPCFC as covariates
Statistical Analysis 2: Comparison: Ligelizumab 120 mg vs Placebo; Test type: Other; p = 0.073, Regression, Logistic; Odds Ratio (OR) = 5.10, 95% CI 2-sided [0.80 to 100.98] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants Who Tolerated a Single Dose of >= 1000 mg (2044 mg Cumulative Tolerated Dose) of Peanut Protein Without Dose-limiting Symptoms at Week 12
Description: Responder rate was defined as the percentage of participants tolerating a single dose of >= 1000 mg (2044 mg cumulative tolerated dose) of peanut protein without dose-limiting symptoms during the double blind placebo controlled food challenge (DBPCFC) conducted at Week 12. The cumulative tolerated dose is the sum of the tolerated doses, not including the reactive dose. Dose-limiting symptoms indicate a true allergic reaction occurring during administration of a single dose of peanut protein at the DBPCFC that should preclude the administration of any further doses in the view of the investigator. Symptoms that require administration of any rescue medication were considered dose-limiting symptoms. Participants with treatment discontinuation or missing more than 1 doses of study drug prior to Week 12 due to reasons other than operational complications caused by public health emergency were considered non-responders.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 47 | 51 | 23
Participants | 14 | 6 | 1
Statistical Analysis 1: Comparison: Ligelizumab 240 mg vs Placebo; Test type: Other; p = 0.018, Regression, Logistic; Odds Ratio (OR) = 9.86, 95% CI 2-sided [1.69 to 188.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ligelizumab 120 mg vs Placebo; Test type: Other; p = 0.164, Regression, Logistic; Odds Ratio (OR) = 3.02, 95% CI 2-sided [0.45 to 59.93] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Who Tolerated a Single Dose of 3000 mg (5044 mg Cumulative Tolerated Dose) of Peanut Protein Without Dose-limiting Symptoms at Week 12
Description: Responder rate was defined as the percentage of participants tolerating a single dose of 3000 mg (5044 mg cumulative tolerated dose) of peanut protein without dose-limiting symptoms during the double blind placebo controlled food challenge (DBPCFC) conducted at Week 12. The cumulative tolerated dose is the sum of the tolerated doses, not including the reactive dose. Dose-limiting symptoms indicate a true allergic reaction occurring during administration of a single dose of peanut protein at the DBPCFC that should preclude the administration of any further doses in the view of the investigator. Symptoms that require administration of any rescue medication were considered dose-limiting symptoms. Participants with treatment discontinuation or missing more than 1 doses of study drug prior to Week 12 due to reasons other than operational complications caused by public health emergency were considered non-responders.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 47 | 51 | 23
Participants | 7 | 5 | 1
Statistical Analysis 1: Comparison: Ligelizumab 240 mg vs Placebo; Test type: Other; p = 0.138, Regression, Logistic; Odds Ratio (OR) = 3.47, 95% CI 2-sided [0.51 to 70.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ligelizumab 120 mg vs Placebo; Test type: Other; p = 0.247, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.30 to 45.56] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Maximum Severity of Symptoms Occurring at Any Challenge Dose of Peanut Protein up to and Including 1000 mg at Week 12
Description: Symptom severity occurring at any challenge dose of peanut protein up to and including 1000 mg during the DBPCFC conducted at Week 12 was categorized as 4 levels: None, Mild, Moderate, Severe. The CoFAR grading system was used to categorize the symptom severity as mild, moderate and severe. Symptom severity for participants who completed DBPCFC without any symptom were categorized as none.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 47 | 51 | 23
Participants
  None | 5 | 2 | 0
  Mild | 15 | 10 | 2
  Moderate | 24 | 37 | 13
  Severe | 3 | 2 | 8
Statistical Analysis 1: Comparison: Ligelizumab 240 mg vs Placebo; Test type: Other; p < 0.001, proportional odds model; Odds Ratio (OR) = 10.59, 95% CI 2-sided [3.63 to 31.56] — proportional odds model adjusting for treatment, age subgroup (12 - 17 yrs, 18 - 55 yrs), log transformed baseline total IgE at screening and region
Statistical Analysis 2: Comparison: Ligelizumab 120 mg vs Placebo; Test type: Other; p = 0.001, proportional odds model; Odds Ratio (OR) = 5.05, 95% CI 2-sided [1.80 to 14.36] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Tolerated a Single Dose of >= 1000 mg (2044 mg Cumulative Tolerated Dose) of Peanut Protein Without Dose-limiting Symptoms at Week 12 After 4 Weeks of Treatment
Description: Responder rate was defined as the percentage of participants tolerating a single dose of >= 1000 mg (2044 mg cumulative tolerated dose) of peanut protein without dose-limiting symptoms during the double blind placebo controlled food challenge (DBPCFC) conducted at Week 12 after 4 weeks of treatment (8 weeks of placebo + 4 weeks of ligelizumab treatment versus 12 weeks of placebo). The cumulative tolerated dose is the sum of the tolerated doses, not including the reactive dose. Participants with treatment discontinuation or missing more than 1 doses of study drug prior to Week 12 due to reasons other than operational complications caused by public health emergency were considered non-responders.
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 46 | 44 | 23
Participants | 8 | 1 | 1
Statistical Analysis 1: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Test type: Other; p = 0.082, Regression, Logistic; Odds Ratio (OR) = 4.73, 95% CI 2-sided [0.74 to 93.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Test type: Other; p = 0.632, Regression, Logistic; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.02 to 16.43] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants Who Tolerated the Specified Peanut Protein Dose Without Dose-limiting Symptoms at Week 52
Description: Responder rate was defined as the percentage of participants tolerating the specified peanut protein doses (>= 600 mg (1044 mg cumulative tolerated dose), >= 1000 mg (2044 mg cumulative tolerated dose) or 3000 mg (5044 mg cumulative tolerated dose)) of peanut protein without dose-limiting symptoms during the double blind placebo controlled food challenge (DBPCFC) conducted at Week 52. The cumulative tolerated dose is the sum of the tolerated doses, not including the reactive dose. Dose-limiting symptoms indicate a true allergic reaction occurring during administration of a single dose of peanut protein at the DBPCFC that should preclude the administration of any further doses in the view of the investigator. Symptoms that require administration of any rescue medication were considered dose-limiting symptoms.
Time Frame: Week 52
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included. Week 52 includes participants who actually reached Week 52 and who reached any week between Week 12 and Week 52 as the end of treatment visit due to study early termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 3 | 2 | 2 | 4 | 0
Participants
  MTD >= 600 mg | 2 | 1 | 0 | 1 |
  MTD >= 1000 mg | 1 | 1 | 0 | 0 |
  MTD = 3000 mg | 1 | 1 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Maximum Tolerated Dose (MTD) of Peanut Protein Without Dose-limiting Symptoms During the DBPCFC at Week 12 and Week 52
Description: Change from baseline in maximum tolerated dose (MTD) of peanut protein without dose-limiting symptoms during the DBPCFC at Week 12 and Week 52. Dose-limiting symptoms indicate a true allergic reaction occurring during administration of a single dose of peanut protein at the DBPCFC that should preclude the administration of any further doses in the view of the investigator.
Time Frame: Baseline, Week 12, Week 52
Population: Full Analysis Set. Only participants with a value at both Baseline and the corresponding post-baseline visit (Week 12 or Week 52) included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 45 | 48 | 46 | 40 | 20
mg
  Week 12 | 274.05 (501.051) | 104.31 (794.248) | 148.98 (754.171) | 44.29 (768.803) | 46.62 (555.207)
  Week 52: number analyzed (Participants) | 3 | 2 | 2 | 4 | 0
  Week 52 | 800.41 (178.687) | 164.23 (459916.375) | 89.55 (408.957) | 146.48 (113.009) |

8. Secondary Outcome: Change From Baseline in Peanut-specific Immunoglobulin E (IgE) at Week 12 and Week 52
Description: Change from baseline of serum levels of peanut-specific immunoglobulin E (IgE)
Time Frame: Baseline, Week 12, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilounits per liter (kU/L)
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 44 | 46 | 45 | 39 | 20
kilounits per liter (kU/L)
  Week 12 | 258.28 (282.477) | 295.60 (321.451) | 302.22 (323.846) | 400.03 (611.676) | -35.52 (179.040)
  Week 52: number analyzed (Participants) | 28 | 26 | 33 | 28 | 18
  Week 52 | 362.36 (436.857) | 297.94 (285.827) | 338.63 (435.532) | 361.44 (587.852) | 174.75 (433.889)

9. Secondary Outcome: Change From Baseline in Peanut-specific Immunoglobulin G4 (IgG4) at Week 12 and Week 52
Description: Change from baseline of serum levels of peanut-specific immunoglobulin G4 (IgG4)
Time Frame: Baseline, Week 12, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 46 | 46 | 45 | 40 | 19
mg/L
  Week 12 | -0.09 (0.65) | 0.35 (3.178) | 0.12 (0.903) | 0.11 (0.789) | 0.03 (0.469)
  Week 52: number analyzed (Participants) | 28 | 27 | 34 | 29 | 17
  Week 52 | -0.01 (0.608) | 0.73 (3.103) | 0.21 (0.909) | 0.01 (0.768) | -0.09 (1.126)

10. Secondary Outcome: Change From Baseline in Skin Prick Test (SPT) Mean Wheal Diameters at Week 16/Week 56
Description: The Skin Prick Test (SPT) is a widely used diagnostic tool for identifying allergen-specific IgE-mediated allergies. During the test, a small amount of allergen, in this case, peanut allergen, is introduced into the skin. The allergen interacts with specific IgE antibodies bound to cutaneous mast cells. This interaction can cause a reaction, resulting in a wheal and flare on the skin. The size of the wheal and flare, specifically the longest diameter and the midpoint orthogonal diameter, were evaluated at each site and the average size of the wheal and flare across all sites was summarized and reported. Considering the study termination, SPT originally scheduled at Week 56 was performed 4 weeks after Week 12 assessment in some patients.
Time Frame: Baseline, Week 16/Week 56
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: undiluted peanut protein (mm)
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 36 | 40 | 37 | 36 | 16
undiluted peanut protein (mm) | -10.85 (6.423) | -8.40 (5.805) | -5.28 (5.237) | -7.25 (7.354) | -2.38 (3.788)
Statistical Analysis 1: Comparison: Ligelizumab 240 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; LS Mean difference = -3.77, 95% CI 2-sided [-5.15 to -2.40] — ANCOVA model with treatment group, age subgroup (12 - 17 years, 18 - 55 years), region, log-transformed baseline total IgE at screening and baseline SPT mean wheal diameter (average dilutions peanut protein) as covariates
Statistical Analysis 2: Comparison: Ligelizumab 120 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; LS Mean difference = -4.93, 95% CI 2-sided [-7.77 to -2.09] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Test type: Other; p = 0.015, ANCOVA; LS Mean difference = -3.20, 95% CI 2-sided [-6.08 to -0.32] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Test type: Other; p = 0.130, ANCOVA; LS Mean difference = -1.68, 95% CI 2-sided [-4.62 to 1.25] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Change From Baseline in Total and Domain Scores in the Food Allergy Quality of Life Questionnaire (FAQLQ) Teenager Form (FAQLQ-TF)
Description: The Food Allergy Quality of Life Questionnaire (FAQLQ) Teenager Form (FAQLQ-TF) is a self-reported instrument designed for adolescents aged 13-17 to assess the impact of food allergy on health-related quality of life (HRQoL). The questionnaire includes three domains (Emotional Impact (EI), Allergen Avoidance and Dietary Restrictions (AADR) and Risk of Accidental Exposure (RAE)). Each item is scored on a 7-point scale (coded as 1-7 in analysis), with a higher score indicating greater impairment in HRQoL. The total score and the domain scores are calculated as the arithmetic average of all completed items. If more than one item in any domain is missing, a domain score should not be calculated for that case. However, a total score could still be calculated if 20% or fewer of the items are missing. Therefore, the range for each item, domain, and the total score is from 1 (minimum) to 7 (maximum). The higher the score, the greater the impairment in HRQoL.
Time Frame: Baseline, Week 12 Part 1 (10 Days Before Day 1 Oral Food Challenge (OFC)), Week 12 Part 2 (3 Days After Day 2 Oral Food Challenge (OFC))
Population: Full Analysis Set. Only adolescent participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 17 | 20 | 15 | 16 | 9
Unit on a scale
  Week 12 Part 1 - Total Score | -0.09 (0.833) | -0.01 (0.779) | -0.30 (0.647) | -0.07 (0.972) | 0.27 (0.835)
  Week 12 Part 2 - Total Score: number analyzed (Participants) | 13 | 17 | 12 | 11 | 8
  Week 12 Part 2 - Total Score | -0.49 (0.839) | -0.13 (0.869) | -0.08 (0.879) | 0.04 (1.255) | 0.09 (0.954)
  Week 12 Part 1 - EI | -0.03 (0.896) | -0.12 (0.846) | -0.40 (0.745) | -0.11 (1.062) | 0.27 (1.034)
  Week 12 Part 2 - EI: number analyzed (Participants) | 13 | 17 | 12 | 11 | 8
  Week 12 Part 2 - EI | -0.51 (1.057) | -0.19 (0.875) | -0.23 (0.737) | -0.05 (1.348) | -0.04 (1.486)
  Week 12 Part 1 - AADR | -0.15 (0.873) | 0.02 (0.977) | -0.35 (0.988) | -0.11 (1.130) | 0.11 (0.599)
  Week 12 Part 2 - AADR: number analyzed (Participants) | 13 | 17 | 12 | 11 | 8
  Week 12 Part 2 - AADR | -0.61 (0.946) | -0.14 (1.004) | -0.08 (1.291) | 0.12 (1.235) | 0.25 (0.628)
  Week 12 Part 1 - RAE | -0.07 (1.085) | 0.08 (0.868) | -0.10 (0.796) | 0.02 (1.016) | 0.54 (1.204)
  Week 12 Part 2 - RAE: number analyzed (Participants) | 13 | 17 | 12 | 11 | 8
  Week 12 Part 2 - RAE | -0.28 (0.718) | -0.04 (1.028) | 0.08 (0.733) | 0.03 (1.366) | -0.04 (1.253)
Statistical Analysis 1: Comparison: Ligelizumab 240 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.173, ANCOVA; LS Mean difference = -0.33, 95% CI 2-sided [-1.03 to 0.36] — ANCOVA with treatment group, baseline PRO scores (FAQLQ) and region as fixed effects and log-transformed total IgE at screening as a covariate
Statistical Analysis 2: Comparison: Ligelizumab 120 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.202, ANCOVA; LS Mean difference = -0.29, 95% CI 2-sided [-0.96 to 0.39] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.151, ANCOVA; LS Mean difference = -0.37, 95% CI 2-sided [-1.09 to 0.34] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.264, ANCOVA; LS Mean difference = -0.23, 95% CI 2-sided [-0.94 to 0.49] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Ligelizumab 240 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.123, ANCOVA; LS Mean difference = -0.43, 95% CI 2-sided [-1.16 to 0.30] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Ligelizumab 120 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.258, ANCOVA; LS Mean difference = -0.23, 95% CI 2-sided [-0.94 to 0.47] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.324, ANCOVA; LS Mean difference = -0.17, 95% CI 2-sided [-0.92 to 0.58] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.473, ANCOVA; LS Mean difference = -0.03, 95% CI 2-sided [-0.78 to 0.73] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Change From Baseline in Total and Domain Scores in the Food Allergy Quality of Life Questionnaire (FAQLQ) Adult Form (FAQLQ-AF)
Description: The Food Allergy Quality of Life Questionnaire (FAQLQ) Adult Form (FAQLQ-AF) is a self-reported instrument designed for adults aged 18-55 to assess the impact of food allergy on health-related quality of life (HRQoL). The questionnaire includes four domains (Emotional Impact (EI), Allergen Avoidance and Dietary Restrictions (AADR), Risk of Accidental Exposure (RAE) and Food Allergy Related Health (FAH)). Each item is scored on a 7-point scale (coded as 1-7 in analysis), with a higher score indicating greater impairment in HRQoL. The total score and the domain scores are calculated as the arithmetic average of all completed items. If more than one item in any domain is missing, a domain score should not be calculated for that case. However, a total score could still be calculated if 20% or fewer of the items are missing. Therefore, the range for each item, domain, and the total score is from 1 (minimum) to 7 (maximum). The higher the score, the greater the impairment in HRQoL.
Time Frame: as for outcome 11
Population: Full Analysis Set. Only adult participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 16 | 17 | 19 | 17 | 9
Unit on a scale
  Week 12 Part 1 - Total Score | -0.01 (0.560) | -0.40 (0.439) | -0.20 (0.601) | 0.00 (0.656) | 0.00 (0.330)
  Week 12 Part 2 - Total Score: number analyzed (Participants) | 10 | 11 | 12 | 12 | 5
  Week 12 Part 2 - Total Score | -0.16 (0.742) | -0.55 (0.671) | -0.60 (0.783) | -0.22 (0.727) | -0.14 (0.542)
  Week 12 Part 1 - EI | 0.07 (0.747) | -0.31 (0.838) | -0.35 (0.601) | -0.04 (0.857) | -0.06 (0.358)
  Week 12 Part 2 - EI: number analyzed (Participants) | 10 | 11 | 12 | 12 | 5
  Week 12 Part 2 - EI | -0.11 (0.980) | -0.47 (1.006) | -0.90 (1.027) | -0.26 (0.828) | 0.00 (0.553)
  Week 12 Part 1 - AADR | -0.07 (0.609) | -0.41 (0.526) | -0.31 (0.805) | -0.12 (0.731) | -0.05 (0.508)
  Week 12 Part 2 - AADR: number analyzed (Participants) | 10 | 11 | 12 | 12 | 5
  Week 12 Part 2 - AADR | -0.10 (0.788) | -0.74 (0.585) | -0.70 (1.106) | -0.20 (0.749) | -0.15 (0.532)
  Week 12 Part 1 - RAE | 0.06 (0.647) | -0.40 (0.427) | 0.02 (0.834) | 0.18 (0.794) | 0.10 (0.471)
  Week 12 Part 2 - RAE: number analyzed (Participants) | 10 | 11 | 12 | 12 | 5
  Week 12 Part 2 - RAE | -0.15 (0.750) | -0.31 (0.917) | -0.34 (0.468) | -0.26 (0.821) | -0.33 (0.549)
  Week 12 Part 1 - FAH | -0.17 (1.082) | -0.53 (0.717) | -0.05 (0.788) | 0.06 (1.056) | 0.04 (1.073)
  Week 12 Part 2 - FAH: number analyzed (Participants) | 10 | 11 | 12 | 12 | 5
  Week 12 Part 2 - FAH | -0.47 (0.864) | -0.73 (0.854) | -0.22 (0.770) | -0.06 (1.153) | 0.07 (1.140)
Statistical Analysis 1: Comparison: Ligelizumab 240 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.597, ANCOVA; LS Mean difference = 0.06, 95% CI 2-sided [-0.44 to 0.57] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Ligelizumab 120 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.064, ANCOVA; LS Mean difference = -0.39, 95% CI 2-sided [-0.89 to 0.11] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.191, ANCOVA; LS Mean difference = -0.22, 95% CI 2-sided [-0.72 to 0.28] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.472, ANCOVA; LS Mean difference = -0.02, 95% CI 2-sided [-0.51 to 0.48] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Ligelizumab 240 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.537, ANCOVA; LS Mean difference = 0.03, 95% CI 2-sided [-0.57 to 0.62] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Ligelizumab 120 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.141, ANCOVA; LS Mean difference = -0.32, 95% CI 2-sided [-0.91 to 0.27] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.063, ANCOVA; LS Meand difference = -0.45, 95% CI 2-sided [-1.04 to 0.13] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.368, ANCOVA; LS Mean difference = -0.10, 95% CI 2-sided [-0.68 to 0.48] — [estimate comment as in outcome 11, analysis 1]

13. Secondary Outcome: Change From Baseline in Total Scores in the Food Allergy Independent Measure (FAIM) - Teenager Form (FAIM-TF)
Description: The Food Allergy Independent Measure (FAIM) - Teenager Form (FAIM-TF) is a self-reported instrument designed for adolescents aged 13-17. It aims to reflect the participant's perceived food allergy severity and food allergy-related risk.
  The questionnaire consists of six questions; The first four questions assess the participant's food allergy expectation outcomes and the remaining two questions reflect aspects of the perceived severity of food allergy. Each question is scored on a 7-point scale (coded as 1-7 in analysis), with a greater score indicating a higher level of perceived risk or chance of adverse events occurring. The total score is calculated as the arithmetic average of all completed items. If less than 80% of the items within the score are complete, the total score is not calculated. Therefore, the range for each item and the total score is from 1 (minimum) to 7 (maximum). The higher the score, the greater the perceived risk or chance of adverse events occurring.
Time Frame: as for outcome 11
Population: Full Analysis Set. Only adolescent participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 17 | 19 | 15 | 14 | 9
Unit on a scale
  Week 12 Part 1 - Total Score | -0.03 (0.751) | -0.11 (0.760) | -0.04 (0.529) | 0.31 (0.989) | 0.19 (0.930)
  Week 12 Part 2 - Total Score: number analyzed (Participants) | 13 | 16 | 12 | 9 | 8
  Week 12 Part 2 - Total Score | -0.31 (0.952) | 0.31 (0.784) | -0.07 (0.524) | 0.39 (1.133) | 0.25 (1.306)
Statistical Analysis 1: Comparison: Ligelizumab 240 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.225, ANCOVA; LS Mean difference = -0.24, 95% CI 2-sided [-0.87 to 0.39] — ANCOVA with treatment group, baseline PRO scores (FAIM) and region as fixed effects and log-transformed total IgE at screening as a covariate
Statistical Analysis 2: Comparison: Ligelizumab 120 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.153, ANCOVA; LS Mean difference = -0.32, 95% CI 2-sided [-0.93 to 0.30] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.179, ANCOVA; LS Mean difference = -0.30, 95% CI 2-sided [-0.95 to 0.34] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.631, ANCOVA; LS Mean difference = 0.11, 95% CI 2-sided [-0.55 to 0.77] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Ligelizumab 240 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.060, ANCOVA; LS Mean difference = -0.52, 95% CI 2-sided [-1.18 to 0.14] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Ligelizumab 120 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.404, ANCOVA; LS Mean difference = -0.08, 95% CI 2-sided [-0.72 to 0.56] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.135, ANCOVA; LS Mean difference = -0.38, 95% CI 2-sided [-1.06 to 0.30] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.514, ANCOVA; LS Mean difference = 0.01, 95% CI 2-sided [-0.70 to 0.72] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Change From Baseline in Total Scores in the Food Allergy Independent Measure (FAIM) - Adult Form (FAIM-AF)
Description: The Food Allergy Independent Measure (FAIM) - Adult Form (FAIM-AF) is a self-reported instrument designed for adults aged 18-55. It aims to reflect the participant's perceived food allergy severity and food allergy-related risk.
  The questionnaire consists of six questions; The first four questions assess the participant's food allergy expectation outcomes and the remaining two questions reflect aspects of the perceived severity of food allergy. Each question is scored on a 7-point scale (coded as 1-7 in analysis), with a greater score indicating a higher level of perceived risk or chance of adverse events occurring. The total score is calculated as the arithmetic average of all completed items. If less than 80% of the items within the score are complete, the total score is calculated. Therefore, the range for each item and the total score is from 1 (minimum) to 7 (maximum). The higher the score, the greater the perceived risk or chance of adverse events occurring.
Time Frame: as for outcome 11
Population: Full Analysis Set. Only adult participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 16 | 17 | 16 | 17 | 8
Unit on a scale
  Week 12 Part 1 - Total Score | 0.17 (0.574) | -0.23 (0.496) | -0.09 (0.694) | 0.00 (0.489) | 0.17 (0.309)
  Week 12 Part 2 - Total Score: number analyzed (Participants) | 10 | 11 | 10 | 12 | 5
  Week 12 Part 2 - Total Score | -0.23 (0.681) | -0.36 (0.562) | -0.27 (0.492) | -0.24 (0.479) | 0.07 (0.703)
Statistical Analysis 1: Comparison: Ligelizumab 240 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.574, ANCOVA; LS Mean difference = 0.04, 95% CI 2-sided [-0.42 to 0.51] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Ligelizumab 120 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.056, ANCOVA; LS Mean difference = -0.37, 95% CI 2-sided [-0.83 to 0.09] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.069, ANCOVA; LS Mean difference = -0.36, 95% CI 2-sided [-0.83 to 0.12] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Week 12 Part 1 - Total Score; Test type: Other; p = 0.205, ANCOVA; LS Mean difference = -0.19, 95% CI 2-sided [-0.65 to 0.27] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Ligelizumab 240 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.248, ANCOVA; LS Mean difference = -0.20, 95% CI 2-sided [-0.76 to 0.37] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Ligelizumab 120 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.071, ANCOVA; LS Mean difference = -0.42, 95% CI 2-sided [-0.98 to 0.14] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: Placebo 8 Weeks and Ligelizumab 240 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.048, ANCOVA; LS Mean difference = -0.49, 95% CI 2-sided [-1.06 to 0.09] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Placebo 8 Weeks and Ligelizumab 120 mg vs Placebo; Week 12 Part 2 - Total Score; Test type: Other; p = 0.142, ANCOVA; LS Mean difference = -0.30, 95% CI 2-sided [-0.85 to 0.25] — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Change From Baseline in the SF-36v2 Physical Component Score (PCS) and Mental Component Score (MCS)
Description: The SF-36v2 Health Survey is a 36-item instrument that measures generic health-related quality of life. It is designed for use in surveys of general and specific populations, health policy evaluations and clinical practice and research. It contains 8 scales and 2 component summary indices evaluating physical, social and emotional functioning in addition to general health perceptions and mental health. Responses to items allow for direct calculation of scale scores, while the physical component summary (PCS) and mental component summary (MCS) scores are computed from weighted scale scores. For all scales and summary measures, higher scores indicate better health outcomes (PCS and MCS scores range 0 to 100).
Time Frame: Baseline, Week 12 Part 2 (3 Days After Day 2 Oral Food Challenge (OFC))
Population: Full Analysis Set. Only participants with a value at both Baseline and post-baseline visit included.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Ligelizumab 240 mg | Ligelizumab 120 mg | Placebo 8 Weeks and Ligelizumab 240 mg | Placebo 8 Weeks and Ligelizumab 120 mg | Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 12 | 5
Unit on a scale
  Physical Component Score | 0.51 (8.022) | 0.38 (2.912) | 2.13 (3.909) | -2.19 (5.090) | 3.15 (5.342)
  Mental Component Score | -0.15 (9.950) | -0.12 (8.175) | -1.78 (8.458) | -3.26 (8.256) | -9.43 (14.662)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to 30 days after last dose of study medication, up to approximately 22 months.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up.
Groups:
- Placebo Controlled Period (Up to Week 8) Ligelizumab 240 mg SCq4w: Placebo controlled period (Up to Week 8) Ligelizumab 240 mg SCq4w
- Placebo Controlled Period (Up to Week 8) Ligelizumab 120 mg SCq4w: Placebo controlled period (Up to Week 8) Ligelizumab 120 mg SCq4w
- Placebo Controlled Period (Up to Week 8): Placebo: Up to Week 8 (before transition to active treatment) for participants randomized to either the 8-week or 16-week Placebo arm
- Placebo Controlled Period (Up to Week 16) Ligelizumab 240 mg SCq4w: Only participants randomized to Ligelizumab 240 mg subcutaneous (SC) every 4 weeks (q4w) without placebo
- Placebo Controlled Period (Up to Week 16) Ligelizumab 120 mg SCq4w: Only participants randomized to Ligelizumab 120 mg subcutaneous (SC) every 4 weeks (q4w) without placebo
- Placebo Controlled Period (Up to Week 16): Placebo: Up to Week 16 (before transition to active treatment) for participants randomized to the 16-week Placebo arm only
- Any Ligelizumab 240 mg SCq4w (Subcutaneous Injection Every 4 Weeks) - Up to Week 68: Participants randomized to Ligelizumab 240 mg subcutaneous (SC) every 4 weeks (q4w), either with or without Placebo and who took at least one dose of active treatment during the entire study period
- Any Ligelizumab 120 mg SCq4w (Subcutaneous Injection Every 4 Weeks) - Up to Week 68: Participants randomized to Ligelizumab 120 mg subcutaneous (SC) every 4 weeks (q4w), either with or without Placebo and who took at least one dose of active treatment during the entire study period
Arm/Group | Placebo Controlled Period (Up to Week 8) Ligelizumab 240 mg SCq4w | Placebo Controlled Period (Up to Week 8) Ligelizumab 120 mg SCq4w | Placebo Controlled Period (Up to Week 8): Placebo | Placebo Controlled Period (Up to Week 16) Ligelizumab 240 mg SCq4w | Placebo Controlled Period (Up to Week 16) Ligelizumab 120 mg SCq4w | Placebo Controlled Period (Up to Week 16): Placebo | Any Ligelizumab 240 mg SCq4w (Subcutaneous Injection Every 4 Weeks) - Up to Week 68 | Any Ligelizumab 120 mg SCq4w (Subcutaneous Injection Every 4 Weeks) - Up to Week 68
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/51 | 0/113 | 0/47 | 0/51 | 0/23 | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/51 | 0/113 | 0/47 | 0/51 | 0/23 | 0/99 | 1/101
Other Adverse Events (participants affected / at risk) | 21/47 | 17/51 | 27/113 | 26/47 | 20/51 | 9/23 | 57/99 | 53/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Controlled Period (Up to Week 8) Ligelizumab 240 mg SCq4w (N=47) | Placebo Controlled Period (Up to Week 8) Ligelizumab 120 mg SCq4w (N=51) | Placebo Controlled Period (Up to Week 8): Placebo (N=113) | Placebo Controlled Period (Up to Week 16) Ligelizumab 240 mg SCq4w (N=47) | Placebo Controlled Period (Up to Week 16) Ligelizumab 120 mg SCq4w (N=51) | Placebo Controlled Period (Up to Week 16): Placebo (N=23) | Any Ligelizumab 240 mg SCq4w (Subcutaneous Injection Every 4 Weeks) - Up to Week 68 (N=99) | Any Ligelizumab 120 mg SCq4w (Subcutaneous Injection Every 4 Weeks) - Up to Week 68 (N=101)
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Controlled Period (Up to Week 8) Ligelizumab 240 mg SCq4w (N=47) | Placebo Controlled Period (Up to Week 8) Ligelizumab 120 mg SCq4w (N=51) | Placebo Controlled Period (Up to Week 8): Placebo (N=113) | Placebo Controlled Period (Up to Week 16) Ligelizumab 240 mg SCq4w (N=47) | Placebo Controlled Period (Up to Week 16) Ligelizumab 120 mg SCq4w (N=51) | Placebo Controlled Period (Up to Week 16): Placebo (N=23) | Any Ligelizumab 240 mg SCq4w (Subcutaneous Injection Every 4 Weeks) - Up to Week 68 (N=99) | Any Ligelizumab 120 mg SCq4w (Subcutaneous Injection Every 4 Weeks) - Up to Week 68 (N=101)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 1 | 1
Injection site erythema (General disorders) | 5 | 7 | 0 | 6 | 8 | 0 | 15 | 13
Injection site induration (General disorders) | 3 | 0 | 2 | 3 | 1 | 0 | 9 | 2
Injection site oedema (General disorders) | 3 | 1 | 0 | 4 | 2 | 0 | 7 | 3
Injection site pain (General disorders) | 2 | 3 | 4 | 3 | 3 | 0 | 6 | 4
Injection site pruritus (General disorders) | 3 | 0 | 0 | 3 | 0 | 0 | 4 | 1
Injection site swelling (General disorders) | 2 | 4 | 0 | 2 | 4 | 0 | 6 | 4
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 1
COVID-19 (Infections and infestations) | 1 | 2 | 2 | 5 | 5 | 0 | 7 | 14
Influenza (Infections and infestations) | 1 | 1 | 0 | 2 | 3 | 0 | 5 | 6
Nasopharyngitis (Infections and infestations) | 4 | 2 | 5 | 8 | 3 | 3 | 19 | 14
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 7 | 3 | 4 | 2 | 8 | 9
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 3 | 0 | 0 | 3 | 2
Headache (Nervous system disorders) | 2 | 3 | 5 | 4 | 4 | 1 | 10 | 12
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 4 | 0 | 2 | 7 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 5 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 7 | 1 | 0 | 11 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT04984876/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04984876/SAP_001.pdf